CLINICAL TRIAL: NCT01064817
Title: A Randomized, Double-Masked, Placebo-Controlled Study of PRM-151 in the Prevention of Postoperative Scarring in Glaucoma Patients Following Primary Trabeculectomy
Brief Title: PRM-151 in the Prevention of Scarring Following Trabeculectomy
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Hoffmann-La Roche (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: GA42405; PRM151B-21GL (Other: Promedior, Inc.); 2009-017859-98 (EudraCT Number)
Record Dates: First submitted 2010-02-05; First posted 2010-02-08 (Estimated); Results first posted 2014-08-07 (Estimated); Last update posted 2022-04-28 (Actual); Status verified 2022-03

CONDITIONS: Glaucoma
Keywords: glaucoma, trabeculectomy
MeSH Terms: conditions — Glaucoma | interventions — PRM-151

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- PRM-151 (Experimental): PRM-151 (recombinant human serum amyloid P, recombinant human pentraxin 2)
  Interventions: Drug: PRM-151
- Placebo (Placebo Comparator): Placebo
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: PRM-151 — PRM-151 2 milligrams (mg) (0.1 mL volume) by subconjunctival injection Days 1 (immediately following trabeculectomy), 2, 3, 5 and 9
  Other Names: recombinant human serum amyloid P; recombinant human pentraxin 2
  Arms: PRM-151
Drug: Placebo — Placebo solution (0.1 mL volume) by subconjunctival injection Days 1 (immediately following trabeculectomy), 2, 3, 5 and 9
  Arms: Placebo

SUMMARY:
This study will assess the safety and tolerability of PRM-151 administered as a subconjunctival injection and explore the effect of PRM-151 on various correlates of the wound healing process that occurs in the eye after glaucoma filtration surgery.

DETAILED DESCRIPTION:
Glaucoma is a disease of the eye which affects the optic nerve (the nerve that sends signals from the eye to the brain) and is associated with visual field defects and potential blindness. The treatment of glaucoma involves lowering the pressure in the eye, which is often (but not always) elevated due to accumulation of fluid inside the eye that cannot drain away. In the operation called trabeculectomy (a type of filtration surgery), a small channel is created through the sclera (the white of the eye) to allow accumulated fluid to drain away. Scarring may occur after surgery when, during healing, too much collagen (a type of protein) is deposited in the channel. This causes the channel to seal up and the pressure inside the eye to build up again.

The study will be conducted in patients suffering from glaucoma who are due to undergo trabeculectomy. Patients will be randomized to have either PRM-151 or placebo.

ELIGIBILITY:
Inclusion Criteria:

* Men or women of nonchildbearing potential (WONCBP) aged 18 years and older at screening.
* Diagnosis of chronic angle-closure glaucoma or open-angle glaucoma, phakic or pseudophakic, with visual field or optic disc changes characteristic of glaucoma. For pseudophakic glaucoma patients, the cataract surgery performed was with phacoemulsification and through a corneal incision.
* Suitable candidate for trabeculectomy in the study eye which the physician deems as medically necessary.

Exclusion Criteria:

* Diagnosis of glaucoma other than chronic angle-closure glaucoma or open-angle glaucoma (ie., uveitic, traumatic or neovascular glaucoma).
* Any previous ocular surgeries in the study eye involving the upper conjunctiva and sclera.
* History of laser surgeries in the study eye within 90 days before day 1.
* Presence or history of any disease that could affect wound healing.
* Any asymmetric abnormality of the anterior segment which requires additional intervention (surgery or medication).
* Any abnormality other than glaucoma in the study eye that could affect tonometry.
* Presence or history of uveitis within 10 years or any other ocular infection or inflammation within 14 days before day 1.
* Clear corneal phacoemulsification performed within 90 days before day 1.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 124 (Actual)
Dates: Start 2010-06-14 (Actual); Primary Completion 2012-04-30 (Actual); Study Completion 2012-11-14 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Jeffrey Edelson, MD, FRCPC, MHSc, Study Director — Hoffmann-La Roche
Locations (14):
- University Hospital Leuven, Leuven, Belgium
- Czechia (6):
  - Oftalmologicka klinika Brno-Bohunice, Brno
  - Facility Hospital Hradec Kralove, Hradec Králové
  - Palacky University, Olomouc
  - Hospital Pardubice, Pardubice
  - Charles University, Prague
  - Masaryak's Hospital, Ústí nad Labem
- Netherlands (2):
  - UMC St. Radboud West, Nijmegen
  - Eramus Medical Center, Rotterdam
- United Kingdom (5):
  - Cheltenham General Hospital, Gloucestershire
  - St. Thomas, London
  - Norfolk and Norwich University Hospital-NHS Trust, Norwich
  - Oxford Eye Hosiptal, Oxford
  - Royal Hallamshire Hospital, Sheffield

RESULTS

PARTICIPANT FLOW:
Period: All Study Treatment Days 1-9
Arm/Group | PRM-151 | Placebo
Started | 62 | 62
Completed | 62 | 62
Not Completed | 0 | 0
Period: Study Completion
Arm/Group | PRM-151 | Placebo
Started | 62 | 62
Completed | 60 | 62
Not Completed | 2 | 0
Not completed — Physician Decision | 1 | 0
Not completed — Withdrawal by Subject | 1 | 0

BASELINE CHARACTERISTICS:
Population: All subjects screened and enrolled in study
Groups:
- Total: Total of all reporting groups
Arm/Group | PRM-151 | Placebo | Total
Number analyzed (Participants) | 62 | 62 | 124
Age, Continuous [Median (Full Range); unit: years] | 65 [35 to 83] | 68 [39 to 87] | 66 [35 to 87]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 22 | 32 | 54
  Male | 40 | 30 | 70
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 4 | 3 | 7
  White | 58 | 59 | 117
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 3 | 1 | 4
  Not Hispanic or Latino | 59 | 61 | 120
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  Czech Republic | 34 | 39 | 73
  Belgium | 5 | 9 | 14
  Netherlands | 4 | 3 | 7
  United Kingdom | 19 | 11 | 30

OUTCOME MEASURES:

1. Primary Outcome: Safety of Subconjunctival Injection
Description: Number of adverse events (AEs), treatment emergent adverse events (TEAEs), non-ocular TEAEs, Ocular TEAEs, serious adverse events (SAEs), abnormal slit-lamp biomicroscopic findings, and abnormal dilated fundoscopy findings
Time Frame: AEs, slit-lamp, and fundoscopy findings from first injection through end of study; TEAEs from first injection through Day 30
Population: All subjects enrolled in study; all subjects received all study treatment
Measure: Number; unit: Number of occurrences
Arm/Group | PRM-151 | Placebo
Number analyzed (Participants) | 62 | 62
Number of occurrences
  Number of AEs | 274 | 220
  Number of TEAEs | 166 | 113
  Number of Non-ocular TEAEs | 16 | 11
  Number of Ocular TEAEs | 150 | 102
  Number of SAEs | 16 | 7
  Number of abnormal slit-lamp findings | 58 | 108
  Number of abnormal optic nerve findings | 284 | 290
  Number of abnormal retina findings | 18 | 39
  Number of abnormal macula findings | 2 | 4
  Number of abnormal choroid findings | 0 | 1

2. Other Pre Specified Outcome: Successful Intra-ocular Pressure (IOP) Control
Description: Exploratory efficacy outcome measure. Successful IOP control defined as IOP between 6 and 18 mm Hg or 25% reduction from pre-surgical IOP
Time Frame: Day 120
Measure: Number; unit: participants
Arm/Group | PRM-151 | Placebo
Number analyzed (Participants) | 62 | 62
participants | 36 | 46

3. Other Pre Specified Outcome: Bleb Scarring
Description: Exploratory Efficacy Outcome measure: Bleb scarring is graded on a scale from 0-3. 0= none to minimal scarring, 1= mild, 2= moderate, 3= severe scarring.
Time Frame: Day 120
Population: Number of subjects who had assessment of bleb scarring on Day 120
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | PRM-151 | Placebo
Number analyzed (Participants) | 46 | 54
units on a scale | 1.29 (0.663) | 1.30 (0.633)

4. Primary Outcome: Subjects With Safety Related Events or Findings
Description: The number of Subjects with AEs, TEAEs, SAEs, decreased visual acuity, and worsened visual fields
Time Frame: First injection through end of study for AEs, SAEs, visual acuity and visual fields, and from first injection through Day 30 for TEAEs
Measure: Number; unit: participants
Arm/Group | PRM-151 | Placebo
Number analyzed (Participants) | 62 | 62
participants
  Subjects with at least 1 AE | 46 | 47
  Subjects with at least 1 Treatment Emergent AE | 44 | 41
  Subjects with at least 1 SAE | 9 | 6
  Subjects with decreased visual acuity | 0 | 0
  Subjects with worsened visual field | 5 | 5

ADVERSE EVENTS:
Time Frame: SAEs are reported for all subjects from first study treatment injection through end of study (51 weeks). Treatment emergent adverse events are reported as defined in the protocol for all subjects from first study treatment injection through Day 30.
Arm/Group | PRM-151 | Placebo
Serious Adverse Events (participants affected / at risk) | 9/62 | 6/62
Other Adverse Events (participants affected / at risk) | 44/62 | 41/62
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | PRM-151 (N=62) | Placebo (N=62)
Intraocular pressure increased (Investigations) | 2 | 4
Glaucoma (Eye disorders) | 1 | 1
Choroidal detachment (Eye disorders) | 1 | 0
Choroidal effusion (Eye disorders) | 0 | 1
Flat Anterior Chamber of Eye (Eye disorders) | 1 | 0
Retinal vein occlusion (Eye disorders) | 1 | 0
Visual field defect (Nervous system disorders) | 1 | 0
Chronic Lymphocytic Leukaemia (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Rectosigmoid cancer recurrent (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Myocardial infarction (Cardiac disorders) | 1 | 0
Abdominal pain (Gastrointestinal disorders) | 1 | 0
Pancreatitis (Gastrointestinal disorders) | 1 | 0
Vomiting (Gastrointestinal disorders) | 1 | 0
Cerebrovascular disorder (Nervous system disorders) | 1 | 0
Chronic obstructive pulmonary disease (Respiratory, thoracic and mediastinal disorders) | 1 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | PRM-151 (N=62) | Placebo (N=62)
Anterior chamber cell (Eye disorders) | 11 | 11
Conjunctival haemorrhage (Eye disorders) | 10 | 5
Conjunctival hyperemia (Eye disorders) | 9 | 4
Flat anterior chamber of eye (Eye disorders) | 6 | 5
Hyphaema (Eye disorders) | 7 | 3
Anterior chamber flare (Eye disorders) | 6 | 2
Retinal pigmentation (Eye disorders) | 5 | 2
Intraocular pressure increased (Investigations) | 17 | 13

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of 60 days or less